CLINICAL TRIAL: NCT01701973
Title: The Effect of Dipeptidyl Peptidase IV Inhibition on Growth Hormone-Mediated Vasodilation
Brief Title: Effect of DPP4 Inhibition on Growth Hormone Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jessica Koch Devin, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 120078; 1K23HL119602 (NIH)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: obesity; growth hormone
MeSH Terms: conditions — Obesity | interventions — Sitagliptin Phosphate; pegvisomant; Sugars; omega-N-Methylarginine; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (14 healthy subjects) (Other): In Aim 1: Healthy Lean adults are randomized in a double-blinded cross over fashion to sitagliptin versus placebo.
  In Aim 2: Healthy Lean adults receive sitagliptin and are randomized in a double-blinded cross over fashion to pre-treatment with either LNMMA (L-N-Monomethyl-arginine) versus placebo.
  Interventions: Drug: Sitagliptin; Drug: Placebo; Drug: L-NMMA
- Group B (14 healthy subjects) (Other): In Aim 1: Healthy Lean adults are randomized in a double-blinded cross over fashion to sitagliptin versus placebo.
  In Aim 2: Healthy Lean adults receive sitagliptin and are randomized in a double-blinded cross over fashion to pre-treatment with either pegvisomant versus placebo.
  Interventions: Drug: Sitagliptin; Drug: Pegvisomant; Drug: Placebo
- Group C (14 healthy subjects) (Other): In Aim 1: Healthy Lean adults are randomized in a double-blinded cross over fashion to sitagliptin versus placebo.
  In Aim 2: Healthy Lean adults receive sitagliptin and are randomized in a double-blinded cross over fashion to pre-treatment with either Exendin 9-39 versus placebo.
  Interventions: Drug: Sitagliptin; Drug: Placebo; Drug: Exendin 9-39

INTERVENTIONS:
Drug: Sitagliptin — During Aim 1, given on one of two study days (other study day subjects receive placebo.) During Aim 2, given during both of two study days.
  Other Names: Januvia
Drug: Pegvisomant — During Aim 2, given 72 hours prior to one of two study days (Group B subjects only)
  Other Names: Somavert
  Arms: Group B (14 healthy subjects)
Drug: Placebo — During Aim 1, given on one of two study days (other study day subjects receive sitagliptin.) During Aim 2, given on one of two study days (other study day subjects receive either L-NMMA, pegvisomant, or Exendin 9-39 pending their group assignment)
  Other Names: sugar pill
Drug: L-NMMA — During Aim 2, given during one of two study days (Group A subjects only)
  Other Names: L-N-Monomethyl-arginine
  Arms: Group A (14 healthy subjects)
Drug: Exendin 9-39 — During Aim 2, given during one of two study days (Group C subjects only)
  Arms: Group C (14 healthy subjects)

SUMMARY:
This study tests the following hypotheses:

Aim 1: Test the hypothesis that acute dipeptidyl peptidase 4 (DPP4) inhibition with the currently available anti-diabetic drug, sitagliptin, will increase stimulated growth hormone (GH) secretion in healthy lean adults by decreasing the degradation of growth hormone releasing hormone (GHRH).

Aim 2: Test the hypothesis that decreased degradation of GHRH during acute DPP4 inhibition will result in an increase in endothelium-dependent vasodilation mediated by GH and independent from GLP1 (glucagon like peptide-1) in healthy lean adults.

This study promises to provide novel data regarding how this increasingly used class of anti-diabetic drugs affects the pituitary GH axis and could affect blood vessel relaxation. Growth hormone levels are low in the setting of obesity and pre-diabetes. A further study may evaluate the effect of chronic DPP4 inhibitor therapy in a population of patients with obesity and pre-diabetes.

DETAILED DESCRIPTION:
Growth hormone secretion is low in patients with obesity, insulin resistance, and hyperlipidemia. GH therapy in these populations and others has been limited by side effects which include hyperglycemia. Another strategy to increase GH secretion is to enhance pulsatile GH secretion by growth hormone releasing hormone. Growth hormone releasing hormone (GHRH) has a half life of 5 minutes due to its rapid inactivation by DPP4. An alternative strategy to increase endogenous GH secretion is by inhibiting degradation of GHRH by DPP4. DPP4 inhibitors are currently approved therapies for the treatment of hyperglycemia in patients with type 2 diabetes mellitus. They additionally cause blood vessel relaxation. We therefore propose to test the hypothesis that DPP4 inhibition simultaneously enhances GH secretion while improving blood glucoses and vascular function in patient populations with low GH and increased cardiovascular risk. These preliminary aims serve primarily as a novel "proof of concept" study to define the effect of acute pharmacologic DPPIV inhibition on stimulated GH secretion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years inclusive
* BMI ≤ 25 kg/m2
* For female subjects:

Status-post surgical sterilization, or If of child-bearing potential, utilization of a barrier method of birth control following negative serum pregnancy test at screening visit and on every study day

Exclusion Criteria:

* Smoking
* Type 1 or Type 2 Diabetes Mellitus, as defined by a fasting glucose of 126 mg/dL or greater at the time of screening visit or the use of anti-diabetic medication
* Hypertension, as defined by an untreated seated systolic blood pressure (SBP) greater than 140 mmHg and/or an untreated diastolic blood pressure (DBP) greater than 90 mmHg at the time of screening visit or the use of anti-hypertensive medication
* History of reported or recorded hypoglycemia (plasma glucose < 70 mg/dL)
* Pregnancy and/or Breast-Feeding
* Use of any medication other than multivitamin, including use of transdermal as well as oral hormone replacement therapy or use of oral contraceptive therapy
* Anemia defined as hematocrit <35% at screening visit
* Cardiovascular or cerebrovascular disease, including history of myocardial infarction, history of congestive heart failure, history of stroke
* Pulmonary Hypertension
* Abnormal thyroid hormone levels (TSH) at the time of screening visit
* Abnormal serum insulin like growth factor-1 (IGF-1) at the time of screening visit
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m^2
* Impaired hepatic function (alanine or aspartate transaminase > 2 X upper limit of normal range)
* Treatment with an investigational drug in the 1 month preceding the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica K Devin, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Wilson JR, Brown NJ, Nian H, Yu C, Bidlingmaier M, Devin JK. Dipeptidyl Peptidase-4 Inhibition Potentiates Stimulated Growth Hormone Secretion and Vasodilation in Women. J Am Heart Assoc. 2018 Feb 25;7(5):e008000. doi: 10.1161/JAHA.117.008000. PMID 29478970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Lean Adults are randomized to two cross-over studies (Aim 1 and Aim 2).
Pre-assignment Details: In Aim 1, Healthy adults were randomized in a double-blinded cross-over fashion to sitagliptin vs placebo. A minimum 8 week wash-out separated Aims 1 & 2. 23 of the same adults who completed Aim 1 participated in Aim 2. In Aim 2, these adults were divided into three subgroups and randomized to sitagliptin+placebo vs. sitagliptin+antagonist.
Groups:
- Aim 1: Sitagliptin, Then Placebo; Aim 1: Placebo, Then Sitagliptin: In Aim 1: Healthy Lean adults are randomized in a double-blinded cross over fashion to sitagliptin versus placebo.
- Aim 2: Sitagliptin + Placebo,Then Sitagliptin + LNMMA; Aim 2:Sitagliptin + LNMMA, Then Sitagliptin + Placebo: In Aim 2: Healthy Lean adults receive sitagliptin and are randomized in a double-blinded cross over fashion to pre-treatment with either L-NMMA (L-N-Monomethyl-arginine) versus placebo.
- Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Pegvisomant; Aim 2: Sitagliptin + Pegvisomant, Then Sitagliptin + Placebo: In Aim 2: Healthy Lean adults receive sitagliptin and are randomized in a double-blinded cross over fashion to pre-treatment with either pegvisomant versus placebo.
- Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Exendin 9-39; Aim 2: Sitagliptin + Exendin 9-39, Then Sitagliptin + Placebo: In Aim 2: Healthy Lean adults receive sitagliptin and are randomized in a double-blinded cross over fashion to pre-treatment with either Exendin 9-39 versus placebo.
Period: Aim 1: First Intervention (1 Day)
Arm/Group | Aim 1: Sitagliptin, Then Placebo | Aim 1: Placebo, Then Sitagliptin | Aim 2: Sitagliptin + Placebo,Then Sitagliptin + LNMMA | Aim 2:Sitagliptin + LNMMA, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Pegvisomant | Aim 2: Sitagliptin + Pegvisomant, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Exendin 9-39 | Aim 2: Sitagliptin + Exendin 9-39, Then Sitagliptin + Placebo
Started | 23 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 23 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Aim 1: Second Intervention (1 Day)
Arm/Group | Aim 1: Sitagliptin, Then Placebo | Aim 1: Placebo, Then Sitagliptin | Aim 2: Sitagliptin + Placebo,Then Sitagliptin + LNMMA | Aim 2:Sitagliptin + LNMMA, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Pegvisomant | Aim 2: Sitagliptin + Pegvisomant, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Exendin 9-39 | Aim 2: Sitagliptin + Exendin 9-39, Then Sitagliptin + Placebo
Started | 22 (1 subject was lost to follow-up in between Periods 1 and 2.) | 17 (3 subjects were lost to follow-up in between Periods 1 and 2.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 22 | 17 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Aim 2: First Intervention (1 Day)
Arm/Group | Aim 1: Sitagliptin, Then Placebo | Aim 1: Placebo, Then Sitagliptin | Aim 2: Sitagliptin + Placebo,Then Sitagliptin + LNMMA | Aim 2:Sitagliptin + LNMMA, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Pegvisomant | Aim 2: Sitagliptin + Pegvisomant, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Exendin 9-39 | Aim 2: Sitagliptin + Exendin 9-39, Then Sitagliptin + Placebo
Started | 0 | 0 | 5 | 4 | 2 | 3 | 5 | 4
Completed | 0 | 0 | 5 | 4 | 2 | 3 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Aim 2: Second Intervention (1 Day)
Arm/Group | Aim 1: Sitagliptin, Then Placebo | Aim 1: Placebo, Then Sitagliptin | Aim 2: Sitagliptin + Placebo,Then Sitagliptin + LNMMA | Aim 2:Sitagliptin + LNMMA, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Pegvisomant | Aim 2: Sitagliptin + Pegvisomant, Then Sitagliptin + Placebo | Aim 2: Sitagliptin + Placebo, Then Sitagliptin + Exendin 9-39 | Aim 2: Sitagliptin + Exendin 9-39, Then Sitagliptin + Placebo
Started | 0 | 0 | 5 | 4 | 2 | 3 | 5 | 3 (1 subject was lost to follow-up in between Periods 3 and 4.)
Completed | 0 | 0 | 5 | 4 | 2 | 3 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants From All Groups: Data was collected as one group
Arm/Group | Participants From All Groups
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Stimulated Peak Growth Hormone Level
Description: Subjects underwent two study days separated by a washout period. On one study day they will receive sitagliptin and on another placebo, in a randomized double-blind fashion. Growth hormone secretion was stimulated using arginine (30 grams i.v. over 30 minutes) on each study day. Growth hormone levels were assessed during a 3 hour period following arginine stimulation.
Time Frame: Growth Hormone Level at 30 minutes (i.e. at completion of arginine infusion), 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
Population: Data from all subjects who completed both study days in Aim 1 were analyzed. Subjects represented young, healthy adults without any chronic medical conditions and who did not take any medications. Oral birth control use was not permitted.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Aim 1: Sitagliptin,Female Participants; Aim 1: Placebo, Female Participants; Aim 1: Sitagliptin, Male Participants; Aim 1: Placebo, Male Participants: Subjects underwent two study days separated by a washout period. On one study day they received sitagliptin and on another placebo, in a randomized double-blind fashion. Growth hormone secretion was stimulated using arginine on each study day. Growth hormone levels were assessed during a 3 hour period following arginine stimulation.
Arm/Group | Aim 1: Sitagliptin,Female Participants | Aim 1: Placebo, Female Participants | Aim 1: Sitagliptin, Male Participants | Aim 1: Placebo, Male Participants
Number analyzed (Participants) | 29 | 29 | 10 | 10
ng/ml
  30 minutes | 5.2 (4.2) | 3.1 (3.3) | 1.9 (1.9) | 2.0 (2.3)
  45 minutes | 9.5 (6.1) | 6.6 (5.0) | 3.4 (3.5) | 3.9 (3.3)
  60 minutes | 9.4 (6.4) | 7.0 (6.0) | 3.0 (3.6) | 3.3 (2.3)
  90 minutes | 5.0 (3.4) | 6.4 (4.8) | 1.1 (1.00) | 2.1 (2.0)
  120 minutes | 2.7 (2.1) | 4.2 (3.4) | 1.5 (3.1) | 0.9 (0.8)
  150 minutes | 1.8 (2.5) | 2.4 (2.1) | 2.2 (4.3) | 1.8 (3.3)
  180 minutes | 0.9 (0.9) | 1.3 (1.9) | 1.0 (1.9) | 1.0 (1.8)

2. Primary Outcome: Aim 1: Percent Change From Baseline in Forearm Vascular Resistance
Description: Forearm blood flow was determined by strain gauge plethysmography. Forearm vascular resistance was then calculated by dividing this into mean arterial pressure. The percent change from baseline was determined at each timepoint.
Time Frame: Percent change from baseline in forearm vascular resistance at 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Aim 1: Sitagliptin,Female Participants; Aim 1: Placebo, Female Participants; Aim 1: Sitagliptin, Male Participants; Aim 1: Placebo, Male Participants: Subjects underwent two study days separated by a washout period. On one study day they received sitagliptin and on another placebo, in a randomized double-blind fashion. Growth hormone secretion was stimulated using arginine on each study day. Forearm vascular resistance (FVR) was assessed during a 3 hour period following arginine stimulation.
Arm/Group | Aim 1: Sitagliptin,Female Participants | Aim 1: Placebo, Female Participants | Aim 1: Sitagliptin, Male Participants | Aim 1: Placebo, Male Participants
Number analyzed (Participants) | 29 | 29 | 10 | 10
percentage change from baseline
  30 minutes | -5.0677 (18.56794) | -5.3498 (19.60881) | 1.4929 (21.57596) | -11.2235 (13.60628)
  60 minutes | -5.1365 (16.61555) | -1.0195 (22.62776) | 6.7355 (23.96889) | 4.6875 (31.77169)
  90 minutes | -10.1867 (22.00489) | -1.6694 (31.84989) | 1.0144 (28.50393) | -3.8029 (35.33295)
  120 minutes | -12.5192 (31.29272) | -5.0763 (26.06546) | -10.3674 (32.22945) | -2.7449 (31.52281)
  150 minutes | -24.1962 (23.92090) | -11.8335 (27.88447) | -9.7129 (30.40280) | -7.1590 (30.41909)
  180 minutes | -22.4043 (27.60020) | -16.5358 (32.22119) | -11.9609 (20.50786) | -15.0591 (25.33331)

3. Primary Outcome: Aim 1: Percent Change From Baseline in Forearm Blood Flow
Description: Forearm blood flow was determined by strain gauge plethysmography. The percent change from baseline was determined at each timepoint.
Time Frame: Percent change from baseline in forearm blood flow at 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Aim 1: Sitagliptin,Female Participants; Aim 1: Placebo, Female Participants; Aim 1: Sitagliptin, Male Participants; Aim 1: Placebo, Male Participants: Subjects underwent two study days separated by a washout period. On one study day they received sitagliptin and on another placebo, in a randomized double-blind fashion. Growth hormone secretion was stimulated using arginine on each study day. Forearm blood flow was assessed during a 3 hour period following arginine stimulation.
Arm/Group | Aim 1: Sitagliptin,Female Participants | Aim 1: Placebo, Female Participants | Aim 1: Sitagliptin, Male Participants | Aim 1: Placebo, Male Participants
Number analyzed (Participants) | 29 | 29 | 10 | 10
percent change from baseline
  30 minutes | 0.4835 (19.44436) | 1.6458 (19.42502) | -.0238 (23.86278) | 9.2597 (14.60368)
  60 minutes | 5.3416 (21.33943) | 4.9101 (37.42841) | -2.8869 (25.79685) | 0.6789 (24.91588)
  90 minutes | 15.9192 (36.11077) | 11.7285 (47.44341) | 1.5212 (30.57639) | 13.5358 (37.76659)
  120 minutes | 23.2248 (40.83970) | 10.3081 (28.31870) | 20.1185 (38.89402) | 9.9379 (28.93967)
  150 minutes | 39.9269 (45.00577) | 19.7355 (30.90766) | 21.6011 (42.67343) | 15.0944 (34.56449)
  180 minutes | 40.6354 (50.48606) | 30.0924 (36.51124) | 16.8489 (24.95539) | 26.1772 (34.75120)

4. Primary Outcome: Aim 2: Percent Change From Baseline in Forearm Blood Flow
Description: Subjects undergo two study days separated by a washout period. On one study day they received sitagliptin plus another study drug and on another sitagliptin plus placebo, in a randomized double-blind fashion. Forearm blood flow was assessed at each visit.
Time Frame: as for outcome 3
Population: 19 of the original 29 females in Aim 1 returned to complete two more study days (Aim 2) in which they received sitagliptin + double-blinded study drug vs. sitagliptin plus placebo in a cross-over study. Three men from Aim 1 also returned to complete two more study days (Aim 2).
Measure: Mean (Standard Error); unit: percent change from baseline
Groups:
- Aim 2: Sitagliptin and LNMMA, Female Participants; Aim 2: Sitagliptin and Placebo, Females in LNMMA Group: Seven of the original 29 women returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus L-N-monomethylarginine (LNMMA) and on another sitagliptin plus placebo, in a randomized cross-over fashion.
- Aim 2: Sitagliptin and LNMMA, Male Participants; Aim 2: Sitagliptin and Placebo, Males in LNMMA Group: Two of the men in Aim 1 returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus L-N-monomethylarginine (LNMMA) and on another sitagliptin plus placebo, in a randomized cross-over fashion.
- Aim 2: Sitagliptin and Pegvisomant, Female Participants; Aim 2: Sitagliptin & Placebo, Females in Pegvisomant Group: Five of the original 29 women returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus pegvisomant and on another sitagliptin plus placebo, in a randomized cross-over fashion. The protocol specified a priori not to study men further if the first seven men randomized to sitagliptin vs. placebo in Aim 1 showed no effect of sitagliptin in men.
- Aim 2: Sitagliptin and Exendin 9-39, Female Participants; Aim 2: Sitagliptin and Placebo, Females in Exendin 9-39 Group: Seven of the original 29 women returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus Exendin 9-39 and on another sitagliptin plus placebo, in a randomized cross-over fashion.
- Aim 2: Sitagliptin and Exendin 9-39, Male Participant; Aim 2: Sitagliptin and Placebo, Male in Exendin 9-39 Group: One of the men from Aim 1 returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus Exendin 9-39 and on another sitagliptin plus placebo, in a randomized cross-over fashion.
Arm/Group | Aim 2: Sitagliptin and LNMMA, Female Participants | Aim 2: Sitagliptin and Placebo, Females in LNMMA Group | Aim 2: Sitagliptin and LNMMA, Male Participants | Aim 2: Sitagliptin and Placebo, Males in LNMMA Group | Aim 2: Sitagliptin and Pegvisomant, Female Participants | Aim 2: Sitagliptin & Placebo, Females in Pegvisomant Group | Aim 2: Sitagliptin and Exendin 9-39, Female Participants | Aim 2: Sitagliptin and Placebo, Females in Exendin 9-39 Group | Aim 2: Sitagliptin and Exendin 9-39, Male Participant | Aim 2: Sitagliptin and Placebo, Male in Exendin 9-39 Group
Number analyzed (Participants) | 7 | 7 | 2 | 2 | 5 | 5 | 7 | 7 | 1 | 1
percent change from baseline
  30 minutes | -0.71 (6.75) | -9.34 (8.60) | 5.17 (4.27) | 14.78 (14.78) | 15.64 (5.06) | 0.39 (8.93) | -7.33 (8.66) | -0.98 (12.08) | -7.59 (NA) — Cannot be determined with 1 participant. | -22.67 (NA) — Cannot be determined with 1 participant.
  60 minutes | -3.64 (12.68) | -17.06 (12.93) | 7.05 (4.06) | 4.56 (0.97) | 6.58 (10.16) | 16.10 (12.79) | -10.54 (8.53) | 6.95 (9.53) | 9.37 (NA) — Cannot be determined with 1 participant. | -13.00 (NA) — Cannot be determined with 1 participant.
  90 minutes | 3.24 (10.02) | -6.35 (16.60) | 25.69 (6.25) | 20.32 (12.83) | 36.96 (14.71) | 16.67 (33.39) | 2.23 (8.69) | 2.08 (11.60) | 5.36 (NA) — Cannot be determined with 1 participant. | -18.33 (NA) — Cannot be determined with 1 participant.
  120 minutes | 4.22 (12.54) | 9.80 (18.23) | 32.92 (0.97) | 56.26 (55.06) | 54.10 (21.87) | 41.97 (31.29) | 31.10 (9.04) | 22.24 (11.14) | 16.52 (NA) — Cannot be determined with 1 participant. | -22.00 (NA) — Cannot be determined with 1 participant.
  150 minutes | 16.09 (13.00) | 11.26 (28.45) | 26.27 (13.73) | 71.51 (76.00) | 59.08 (32.36) | 26.87 (17.56) | 29.48 (8.22) | 15.59 (8.26) | 45.98 (NA) — Cannot be determined with 1 participant. | 1.33 (NA) — Cannot be determined with 1 participant.
  180 minutes | 14.80 (15.85) | 17.12 (20.53) | 29.24 (35.21) | 65.31 (80.28) | 51.21 (26.07) | 43.51 (26.31) | 30.76 (8.88) | 27.11 (12.21) | 54.91 (NA) — Cannot be determined with 1 participant. | -1.67 (NA) — Cannot be determined with 1 participant.

5. Primary Outcome: Aim 2: Percent Change From Baseline in Forearm Vascular Resistance
Description: Subjects undergo two study days separated by a washout period. On one study day they will receive sitagliptin plus another study drug and on another sitagliptin plus placebo, in a randomized double-blind fashion. Forearm blood flow was assessed at each visit every 30 minutes for 3 hours. This was divided into mean arterial pressure to determine forearm vascular resistance.
Time Frame: as for outcome 2
Population: 19 of the original 29 females who participated in Aim 1 returned to complete an additional two study days (Aim 2) in which they received sitagliptin + double-blinded study drug vs. sitagliptin plus placebo in a cross-over study. Three men from Aim 1 also returned to complete two more study days (Aim 2).
Measure: Mean (Standard Error); unit: percent change from baseline
Groups:
- Aim 2: Sitagliptin and LNMMA, Female Participants; Aim 2: Sitagliptin and Placebo, Females in LNMMA Group: Seven of the original 29 women returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus LNMMA and on another sitagliptin plus placebo, in a randomized cross-over fashion.
- Aim 2: Sitagliptin & Placebo,Females in Pegvisomant Group: Five of the original 29 women returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus pegvisomant and on another sitagliptin plus placebo, in a randomized cross-over fashion. The protocol specified a priori not to study men further if the first seven men randomized to sitagliptin vs. placebo in Aim 1 showed no effect of sitagliptin in men.
- Aim 2: Sitagliptin and Exendin 9-39, Male Participant; Aim 2: Sitagliptin and Placebo, Male in Exendin 9-39 Group: One of the men in Aim 1 returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus Exendin 9-39 and on another sitagliptin plus placebo, in a randomized cross-over fashion.
Arm/Group | Aim 2: Sitagliptin and LNMMA, Female Participants | Aim 2: Sitagliptin and Placebo, Females in LNMMA Group | Aim 2: Sitagliptin and LNMMA, Male Participants | Aim 2: Sitagliptin and Placebo, Males in LNMMA Group | Aim 2: Sitagliptin and Pegvisomant, Female Participants | Aim 2: Sitagliptin & Placebo,Females in Pegvisomant Group | Aim 2: Sitagliptin and Exendin 9-39, Female Participants | Aim 2: Sitagliptin and Placebo, Females in Exendin 9-39 Group | Aim 2: Sitagliptin and Exendin 9-39, Male Participant | Aim 2: Sitagliptin and Placebo, Male in Exendin 9-39 Group
Number analyzed (Participants) | 7 | 7 | 2 | 2 | 5 | 5 | 7 | 7 | 1 | 1
percent change from baseline
  30 minutes | -8.67 (9.66) | 8.98 (12.07) | -9.87 (0.82) | -14.60 (12.22) | -20.00 (3.67) | -3.75 (12.43) | 5.30 (8.19) | 4.53 (12.62) | 0.57 (NA) — Cannot be determined with 1 participant. | 27.77 (NA) — Cannot be determined with 1 participant.
  60 minutes | 8.77 (17.03) | 51.82 (36.73) | -9.75 (2.28) | -2.42 (3.34) | -4.05 (10.67) | -10.97 (11.64) | 14.46 (11.08) | -4.26 (7.26) | -11.80 (NA) — Cannot be determined with 1 participant. | 6.73 (NA) — Cannot be determined with 1 participant.
  90 minutes | -4.89 (8.93) | 39.24 (35.45) | -23.34 (8.00) | -16.75 (4.25) | -25.28 (7.02) | 3.79 (19.09) | 1.76 (8.96) | 4.82 (16.53) | -14.02 (NA) — Cannot be determined with 1 participant. | 22.45 (NA) — Cannot be determined with 1 participant.
  120 minutes | 0.99 (11.00) | 21.98 (35.57) | -24.81 (1.18) | -28.34 (21.27) | -32.39 (8.90) | -14.57 (18.78) | -22.37 (6.11) | -13.16 (10.34) | -16.20 (NA) — Cannot be determined with 1 participant. | 26.68 (NA) — Cannot be determined with 1 participant.
  150 minutes | -13.25 (8.49) | 42.27 (44.03) | -20.62 (6.34) | -32.11 (24.34) | -30.12 (11.10) | -14.25 (13.15) | -20.92 (5.30) | -8.49 (9.03) | -32.30 (NA) — Cannot be determined with 1 participant. | -1.32 (NA) — Cannot be determined with 1 participant.
  180 minutes | -10.25 (10.76) | 5.28 (19.22) | -22.56 (13.90) | -19.52 (37.12) | -25.00 (11.92) | -17.97 (15.66) | -22.58 (5.82) | -16.76 (8.94) | -34.69 (NA) — Cannot be determined with 1 participant. | 1.69 (NA) — Cannot be determined with 1 participant.

6. Secondary Outcome: Aim 1: Venous Blood Sampling for Tissue Plasminogen Activator (TPA) Activity Levels
Description: In Aim 1 subjects underwent two study days separated by a washout period. On one study day they received study drug and on another placebo, in a randomized double-blind fashion. Venous blood samples were obtained at each visit.
Time Frame: baseline and every 30 minutes for 180 minutes
Population: Data from the first 14 subjects (7 men and 7 women) who completed both study days in Aim 1 were analyzed. We do not report tPA results from the remaining participants as the manufacturer changed the tPA assay standard and results were not comparable.
Measure: Mean (Standard Error); unit: IU/ml
Groups:
- Aim 1: Sitagliptin,Female Participants: Subjects undergo two study days separated by a washout period. On one study day they received sitagliptin and on another placebo, in a randomized double-blind fashion. Growth hormone secretion was stimulated using arginine on each study day. tPA levels were assessed during a 3 hour period following arginine stimulation.
- Aim 1: Placebo, Female Participants; Aim 1: Sitagliptin, Male Participants; Aim 1: Placebo, Male Participants: Subjects underwent two study days separated by a washout period. On one study day they received sitagliptin and on another placebo, in a randomized double-blind fashion. Growth hormone secretion was stimulated using arginine on each study day. tPA levels were assessed during a 3 hour period following arginine stimulation.
Arm/Group | Aim 1: Sitagliptin,Female Participants | Aim 1: Placebo, Female Participants | Aim 1: Sitagliptin, Male Participants | Aim 1: Placebo, Male Participants
Number analyzed (Participants) | 7 | 7 | 7 | 7
IU/ml
  Baseline prior to Arginine | 0.30 (0.05) | 0.28 (0.05) | 0.44 (0.14) | 0.22 (0.07)
  30 minutes | 0.40 (0.04) | 0.32 (0.04) | 0.28 (0.08) | 0.25 (0.07)
  45 minutes | 0.43 (0.04) | 0.35 (0.04) | 0.40 (0.10) | 0.32 (0.08)
  60 minutes | 0.40 (0.06) | 0.32 (0.05) | 0.37 (0.09) | 0.34 (0.08)
  90 minutes | 0.39 (0.07) | 0.35 (0.06) | 0.34 (0.09) | 0.27 (0.07)
  120 minutes | 0.40 (0.07) | 0.35 (0.04) | 0.38 (0.12) | 0.28 (0.07)
  150 minutes | 0.44 (0.04) | 0.41 (0.04) | 0.42 (0.12) | 0.37 (0.08)
  180 minutes | 0.55 (0.06) | 0.50 (0.05) | 0.51 (0.12) | 0.45 (0.09)

7. Secondary Outcome: Aim 2: Venous Blood Sampling for Tissue Plasminogen Activator (TPA) Activity Levels
Description: Subjects undergo two study days separated by a washout period. On one study day they received sitagliptin plus pegvisomant and on another sitagliptin plus placebo, in a randomized double-blind fashion. Tissue plasminogen activator activity (tPA) was assessed at each visit.
Time Frame: baseline and every 30 minutes until 180 minutes
Population: Five of the original 29 women returned for two more study days separated by a wash-out. As pre-specified in the protocol, men did not complete this portion of the study. We do not report tPA results from participants who received LNMMA and Exendin 9-39 in this table as the manufacturer changed the tPA assay standard and results were not comparable.
Measure: Mean (Standard Error); unit: IU/ml
Groups:
- Aim 2: Sitagliptin and Placebo, Females in Pegvisomant Group; Aim 2: Sitagliptin and Pegvisomant, Female Participants: Five of the original 29 women returned for an additional two study days separated by a wash-out period. On one study day they received sitagliptin plus pegvisomant and on another sitagliptin plus placebo, in a randomized cross-over fashion.
Arm/Group | Aim 2: Sitagliptin and Placebo, Females in Pegvisomant Group | Aim 2: Sitagliptin and Pegvisomant, Female Participants
Number analyzed (Participants) | 5 | 5
IU/ml
  Baseline prior to Arginine | 0.24 (0.05) | 0.10 (0.03)
  30 minutes | 0.26 (0.04) | 0.15 (0.05)
  45 minutes | 0.33 (0.06) | 0.17 (0.06)
  60 minutes | 0.27 (0.08) | 0.14 (0.04)
  90 minutes | 0.26 (0.07) | 0.16 (0.05)
  120 minutes | 0.28 (0.08) | 0.16 (0.05)
  150 minutes | 0.31 (0.07) | 0.20 (0.05)
  180 minutes | 0.35 (0.06) | 0.23 (0.05)

8. Secondary Outcome: Aim 2: Measurement of Growth Hormone (GH) Levels
Description: Subjects undergo two study days separated by a washout period. On one study day they received sitagliptin plus pegvisomant and on another sitagliptin plus placebo, in a randomized double-blind fashion. Growth hormone secretion following arginine stimulation was assessed at each visit. Growth hormone levels were determined using an assay that is not subject to interference by pegvisomant.
Time Frame: baseline and every 30 minutes until 180 minutes
Population: Five of the original 29 women returned for an additional two study days separated by a wash-out period. As pre-specified in the protocol, men did not complete this portion of the study. We did not measure GH levels in participants who received LNMMA or Exendin 9-39 as these drugs are not known to influence GH secretion.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Aim 2: Sitagliptin and Placebo, Females in Pegvisomant Group | Aim 2: Sitagliptin and Pegvisomant, Female Participants
Number analyzed (Participants) | 5 | 5
ng/mL
  30 minutes | 2.99 (1.60) | 4.27 (2.19)
  60 minutes | 5.92 (2.37) | 7.00 (2.20)
  90 minutes | 6.05 (2.39) | 11.53 (4.67)
  120 minutes | 4.06 (2.18) | 6.17 (1.21)
  150 minutes | 1.83 (0.83) | 4.09 (1.33)
  180 minutes | 1.57 (0.82) | 1.77 (0.32)

ADVERSE EVENTS:
Time Frame: The first subject started drug 2/11/13 and the last completed 2/10/2017. In Aim 1, each subject took oral study drug (placebo vs. sitagliptin). Adverse event data was collected over a one month period for each subject. In Aim 2, each subject took oral sitagliptin and also received a single dose of LNMMA, Exendin 9-39 or Pegvisomant based upon their subgroup assigment. Adverse event data was collected over a 6 week period for each subject.
Groups:
- Sitagliptin; Placebo: Healthy lean adults completed a double blinded cross over study in which they took sitagliptin vs. placebo separated by a wash-out.
- Sitagliptin Plus Pegvisomant: Five women from Aim 1 returned for an additional two study days in which they were randomized to sitagliptin plus placebo vs. sitagliptin plus pre-treatment with pegvisomant.
- Sitagliptin Plus LNMMA: 9 participants from Aim 1 returned for an additional two study days in which they were randomized to sitagliptin plus placebo vs. sitagliptin plus L-N-mono-methylarginine (LNMMA).
- Sitagliptin Plus Exendin 9-39: 8 participants from Aim 1 returned for an additional two study days in which they were randomized to sitagliptin plus placebo vs. sitagliptin plus Exendin 9-39.
Arm/Group | Sitagliptin | Placebo | Sitagliptin Plus Pegvisomant | Sitagliptin Plus LNMMA | Sitagliptin Plus Exendin 9-39
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43 | 0/5 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 0/5 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 7/40 | 1/43 | 2/5 | 0/9 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=40) | Placebo (N=43) | Sitagliptin Plus Pegvisomant (N=5) | Sitagliptin Plus LNMMA (N=9) | Sitagliptin Plus Exendin 9-39 (N=8)
Bruising related to placement of intravenous catheter (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Nasal congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Reflux (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dizziness and paresthesias during arginine infusion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abdominal cramping and diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT01701973/Prot_SAP_000.pdf